CLINICAL TRIAL: NCT02783365
Title: Improving the Management of Chronic Pain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Academy of Family Physicians National Research Network (Network)
Responsible Party: Principal Investigator, Benjamin Crenshaw, Assistant Professor, Family and Community Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004283
Record Dates: First submitted 2016-05-17; First posted 2016-05-26 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention uses photo-elicitation and online group support (via Facebook) to improve patients' overall experience of chronic pain and patient-identified areas of function. This intervention was informed by the Photovoice methodology developed by Wang and Burris (1994). Photovoice participants will utilize cameras that enable them to record issues related to their experiences, and subsequently display them in office visits with their physician or mid-level clinician.
  Interventions: Behavioral: Photo-elicitation and online group support
- Control (No Intervention): Patients in the control practices will receive usual care and will be eligible to participate in the intervention after their participation in the study is completed at 12 months.

INTERVENTIONS:
Behavioral: Photo-elicitation and online group support — See above information.
  Arms: Intervention

SUMMARY:
There are an estimated 100 million Americans with chronic pain. The enormity of the problem at the societal level is staggering, not simply in terms of its sheer prevalence but also the societal costs, including health care expenditures, disability compensation, lost productivity, and lost employment potential. The pharmacological focus in treatment tends to give patients with chronic pain a negative stereotype as many are viewed as drug seeking, or worse, they are perceived to have an imaginary illness. It is argued that these stigmas not only negatively affect the patients' healthcare experience, but also perpetuate maladaptive coping. In addition, it is suggested that reliance on pharmacological approaches have contributed to the rate of overdoses from prescribed opioids. In order to address this burden facing society, patients need opportunities to foster a sense of self-efficacy to manage their pain, as well as improve their healthcare experience by allowing them to dialogue with their clinician openly and freely about their chronic pain, and coping strategies.

This study is designed to explore the impact of an intervention using photo-elicitation (based on Photovoice) and online group support (via Facebook) on participants' overall experience of chronic pain and patient-identified areas of function. Photovoice participants will utilize cameras that enable them to record issues related to their experiences, and subsequently display them. This method serves as an empowering tool to connect participants to key stakeholders in the community, facilitates change and opportunities that otherwise would not be available to marginalized groups.

DETAILED DESCRIPTION:
This is a multi-site study occurring between the University of Missouri, and the American Academy of Family Physicians National Research Network (NRN). The University of Missouri will be responsible for the following:

* Coordinating the approval of initial protocol as well as subsequent amendments.
* Ensure that each site is using the correct version of the protocol.
* Serve as the study contact.
* Participate in the selection of qualified sites for participation (the NRN will be responsible for recruitment and randomization. This process will be overseen by MU).
* Monitor progress and oversee all conduct of the study at participating sites.
* Responsible for the data analysis, reporting, integrity, and accuracy of data.

There will be one protocol document, and each site will utilize this document. The lead site (MU) will develop the informed consent, which includes language that data will be shared with the NRN.

The NRN will be the Institutional Review Board (IRB) of record for the 18 practices recruited to participate within the NRN, and will provide a letter of authorization and final IRB approval to the lead PI (MU).

The study will test if a photo elicitation intervention combined with access to online community support and a chronic pain guideline can improve a 3-item measure of chronic pain [the PEG score: Pain intensity (P), Enjoyment of Life (E), and General Activity (G)] and a patient-identified area of function, compared to a group who receive the guideline alone.

ELIGIBILITY:
Inclusion Criteria:

Patients will need to meet the following criteria in order to participate in the study:

* they must be between the ages of 18-75
* they must have an established care relationship with the practitioner (having had at least two previous visits for chronic pain of at least 6 months' duration)
* they must read and understand English
* they must be willing to sign a consent. Patients must have a device to take pictures (e.g., camera, phone, or tablet) and access to the internet in order to complete REDcap (the online data collection tool we will use to capture quantitative data in order to assess intervention impact), and participate in the online discussions via Facebook.

Exclusion Criteria:

* No terminal illness, and/or a life expectancy of < 1yr.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Change in the score on the 3-item measure of chronic pain (PEG) | Change from baseline to 12 months after enrollment
  The PEG asks 3 questions about (1) severity of pain on average in the past week, (2) how much has pain interfered with your life during the past week, and (3) how much has pain interfered with your general activity.

SECONDARY OUTCOMES:
Change in the score on the Pain Self-Efficacy Questionnaire (PSEQ) | Change from baseline to 12 months after enrollment
  The PSEQ is a 10-item questionnaire asking "how confident you are" in performing activities in the specified areas.
Change in the score on the Chronic Pain Acceptance Questionnaire (CPAQ) | Change from baseline to 12 months after enrollment
  We will use 8 of the 20 questions in the CPAQ, which ask about pain acceptance.
Change in score on a scale measuring the patient-centeredness of an office visit (Stewart et al., 2004) | Change from baseline to 12 months after enrollment
  This scale of patient-centeredness asks 14 questions about how patient-centered the office visit was. We will use a subset of the 14 items.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Crenshaw, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Dept. of Family and Community Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will post de-identified data on an open-access website when the study is completed.